CLINICAL TRIAL: NCT04504994
Title: "Fight-or-flight" Versus "Tend-and-befriend" Response to Behavioral and Pharmacological Interventions in Patients With Borderline Personality Disorder - Part I
Brief Title: Stress & Social Cognition in Borderline Personality Disorder
Acronym: SOKO-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Katja Wingenfeld, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: WI 3396/12-1
Record Dates: First submitted 2020-07-30; First posted 2020-08-07 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- exclusion BPD (Experimental): cyberball exclusion condition - BPD patients
  Interventions: Behavioral: inclusion condition
- over-inclusion BPD (Experimental): cyberball over-inclusion condition - BPD patients
  Interventions: Behavioral: inclusion condition
- exclusion healthy controls (Experimental): cyberball exclusion condition - healthy controls
  Interventions: Behavioral: inclusion condition
- over-inclusion healthy controls (Experimental): cyberball over-inclusion condition - healthy controls
  Interventions: Behavioral: inclusion condition

INTERVENTIONS:
Behavioral: inclusion condition — cyberball game: ex- versus over-inclusion condition

SUMMARY:
The investigators will examine whether perceived social exclusion provoke a reduction in prosocial behavior in BPD patients.

DETAILED DESCRIPTION:
The investigators will examine whether perceived social exclusion provoke a reduction in prosocial behavior, such as empathy, in BPD patients and whether this "fight-or-flight" pattern is also seen in other relevant aspects of social behavior, such as sharing and punishment behavior. To induce social exclusion all participants will play cyberball, either the exclusion condition or the (over)inclusion condition before testing

ELIGIBILITY:
Inclusion Criteria:

female patients with BPD and healthy control women, matched for age, body mass index, and education

Exclusion Criteria:

physical illness

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female only
Enrollment: 196 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
empathy | 30 minutes after cyberball
  Multifaceted Empathy Test

SECONDARY OUTCOMES:
sharing behavior: amount of monetary units (max 30) shared with co-player | directly after cyberball
  Computer game

OTHER OUTCOMES:
punishment behavior: number of accepted offers from co-player | 15 minutes after cyberball
  Computer game

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided